CLINICAL TRIAL: NCT02153541
Title: Assessing the Efficacy of Antipyrine Benzocaine Otic Solution in the Ear Canal to Decrease Usage of Rescue Inhalers in Moderate to Severe Asthmatic Adults.
Brief Title: Assessing the Efficacy of CREWS01 to Decrease Usage of Rescue Inhalers in Moderate to Severe Asthmatic Adults
Acronym: CREWS01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Global United Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CREWS01
Record Dates: First submitted 2014-05-21; First posted 2014-06-03 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Glycerol; Oxyquinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glycerin with Oxyquinoline Sulfate (Placebo Comparator): For those participants who receive glycerin with oxyquinoline sulfate placebo, we do not anticipate any change in the usage of rescue inhalers, spirometer scores, asthma diaries, and expired fractionated nitrous oxide levels.
  Interventions: Other: Glycerin with Oxyquinoline Sulfate
- Antipyrine-benzocaine otic solution (Active Comparator): Will be used on 50% of participants, we anticipate reduction in the usage of rescue inhalers, spirometer scores, asthma diaries, and expired fractionated nitrous oxide levels.
  Interventions: Drug: Antipyrine-benzocaine otic solution

INTERVENTIONS:
Drug: Antipyrine-benzocaine otic solution — Participants receiving antipyrine-benzocaine otic solution are expected to decrease usage of rescue inhalers.
  Arms: Antipyrine-benzocaine otic solution
Other: Glycerin with Oxyquinoline Sulfate — 50% of participants will receive the glycerin with oxyquinoline sulfate. These participants will be randomly selected and unaware that they are receiving the placebo and are expected to have no change in usage of rescue inhalers.
  Arms: Glycerin with Oxyquinoline Sulfate

SUMMARY:
This is a double-blind, randomized, placebo-controlled, proof of concept, study in adults with poorly controlled moderate to severe asthma. The researchers believe that by using a local anesthetic to block a certain nerve in the ear, it will improve all aspects of asthma, such as decreasing the numbers of times patients have to use a rescue inhaler, and improving asthma treatment assessment questionnaire scores, with no bad changes to lung function and inflammation.

DETAILED DESCRIPTION:
The proposed four-week, double-blind, placebo controlled study is designed to test the hypothesis that topical auricular anesthesia of the vagus nerve decreases the need for the usage of rescue inhalers in moderate to severe asthma in adults.

We anticipate that up to 50 patients will be enrolled in the trial. Particularly severe risks are not anticipated based on the prior investigational experience with this drug. This trial will be used to generate experience and data to support the design of a larger, crossover, comparator trial investigating the efficacy of antipyrine-benzocaine in reducing the need for rescue inhalers and hospital admissions in moderate to severe asthmatic adults.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe asthma
* Rescue inhaler 3 times per week
* Be able to give informed consent
* Must be on inhaled corticosteroid and long-acting beta agonist (LABA), (either individually or as a combination product) and report using a short-acting beta agonist (SABA) three or more times a week in at least 2 or 3 weeks prior to stud enrollment
* Moderate or severe persistent asthma according to the National Heart, Lung, and Blood Institute (NHLBI) Guidelines, (EPR 2007)
* At least one appointment scheduled with the asthma physician during the 4 weeks of participation.
* Must be able to complete questionnaires over the phone or in person
* Must be able to maintain a basic diary/log of inhaler use and any side effects for 30 days.

Exclusion Criteria:

* Severe psychiatric or cognitive problems
* Known or suspected sensitivity to the investigational medication
* Have a stenotic ear canal
* Have a perforated ear drum
* Active Otitis Media, Otitis Externa, or Mastoiditis
* Allergic to Benzocaine
* Unable to communicate in English
* Any other significant cardiopulmonary disease
* Smokers
* Hospitalized in the last 6 months for pneumonia
* Long term or lingering side effects to COVID19
* Lack of telephone or mobile phone
* Subjects who have received any investigational drug for asthma in the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of CREWS01 (topical auricular anesthesia of the vagus nerve) to decrease usage of rescue inhalers in moderate to severe asthmatic adults Change in usage of rescue inhalers in moderate to severe asthmatic adults in four weeks | Each participant is studied for four weeks
  We anticipate 50% of patients that receive the active ingredient will decrease the usage of rescue inhalers by 50%. If the test of the two-factor interaction in the repeated measures mixed model analysis is statistically significant, and the magnitude of the change in the Crews group is at least 50%, the Crews Maneuver will be considered effective.

SECONDARY OUTCOMES:
Improvement of spirometry scores in moderate to severe asthmatic adults | Each participant is studied for four weeks
  We anticipate 50% of patients that receive the active ingredient will not show a significant decline in spirometry scores and eNO results that do not show a significant increase in subjects on the active drug compared to the placebo, and improvement in both ACT and ATAQ scores of at least 25% over the 4 weeks of study.

OTHER OUTCOMES:
Evaluate the safety of using topical anesthetics in moderate to severe asthmatic adults | Each participant is studied for four weeks
  We anticipate the active medication is safe for topical usage in moderate to severe asthmatic adults. The common side effects of topical anesthetics include, but are not limited to, stinging, burning or itching of the ear canal.

CONTACTS AND LOCATIONS:
Overall Officials: John D Prosser, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing after phase 3 clinical trial completed
Supporting Information: CSR
Time Frame: 6 months after completion of phase 3 clinical trial
Access Criteria: undetermined